CLINICAL TRIAL: NCT00698945
Title: Randomized, Investigator Masked Comparison of Istalol™ 0.5% QD (Timolol Maleate/Sorbitol Complex, ISTA Pharmaceutical) to Brimonidine Tartrate 0.1% BID as Adjunctive Therapy to Latanoprost 0.005% in Adults With Ocular Hypertension (OHT) or Open-Angle Glaucoma (OAG)
Brief Title: Comparison of Istalol™ 0.5% QD (Timolol Maleate/Sorbitol Complex, ISTA Pharmaceutical) to Brimonidine Tartrate 0.1% BID as Adjunctive Therapy to Latanoprost 0.005% in Adults With Ocular Hypertension (OHT) or Open-Angle Glaucoma (OAG)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Dr. Bacharach, North Bay Eye Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5358
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Timolol; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 2 (Active Comparator): Alphagan
  Interventions: Drug: Alphagan
- 1 (Active Comparator): Istalol and Optive
  Interventions: Drug: Istalol and Optive

INTERVENTIONS:
Drug: Istalol and Optive — Istalol: one drop a day for 28 days Optive: one drop a day for 28 days
  Arms: 1
Drug: Alphagan — Alphagan: two drops a day for 28 days
  Arms: 2

SUMMARY:
To assess the additional benefit of common adjunctive classes on the diurnal IOP curve in patients assessed as needing additional treatment to reach target intraocular pressure (IOP). To demonstrate superiority of IOP control with Istalol 0.5% QD compared to Brimonidine Tartrate 0.2% BID as adjunctive therapy in adults with uncontrolled IOP's (determined by P.I. based on target pressures) currently treated with Latanoprost 0.05% in the study eye(s).

ELIGIBILITY:
Inclusion Criteria:

1. Patients, male or female of any race or ethnicity, 18 years of age or older, diagnosed with ocular hypertension or open-angle glaucoma (with or without pseudoexfoliative or pigmentary dispersion component).
2. Stable use of Latanoprost 0.005% for a minimum of 30 days prior to screening visit.
3. VA of 20/200 or better in either eye
4. Pachymetry of 600 microns or less
5. Visual Field within 6 months of screening visit
6. Patients who use contact lenses are allowed to participate provided that they will remove lenses 15 minutes before dosing
7. Patients who satisfy all informed consent requirements may be included in the study.

Exclusion Criteria:

1. Females of childbearing potential (those who are not surgically sterile, postmenopausal or using a reliable birth control method) will be excluded from the study.
2. Any allergic component or contraindication to the study medications
3. Pachymetry of 600 microns or greater
4. Systemic corticosteroids not on a stable regimen within 30 days of screening visit.
5. Any concurrent topical agents that can not be discontinued during the course of the trial (natural tears are acceptable)
6. Significant ocular surface abnormalities
7. Patients with any form of glaucoma other than ocular hypertension or open-angle glaucoma
8. Patients who have been on an investigational therapy within 30 days prior to screening visit
9. History of ocular trauma within the past 3 months
10. Intraocular surgery within the past 3 months
11. Ocular laser surgery within the past 3 months
12. Any abnormality preventing reliable applanation tonometry of either eye
13. VA of 20/200 or greater in either eye
14. History or evidence of clinically significant illness or conditions which would make the patient, in the opinion of the investigator, not suitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Trough and peak intraocular pressure | 2-4 months

SECONDARY OUTCOMES:
Tolerability of study medication | 2-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bacharach, M.D, Principal Investigator — North Bay Eye Associates,Inc.
Locations (1):
- North Bay Eye Associates, Inc., Petaluma, California, United States